CLINICAL TRIAL: NCT03622905
Title: ADvance II: A 12-month Double-blind, Randomized, Controlled Study to Evaluate the Safety and Efficacy of Deep Brain Stimulation of the Fornix (DBS-f) in Patients With Mild Probable Alzheimer's Disease
Brief Title: ADvance II Study: DBS-f in Patients With Mild Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Functional Neuromodulation Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FNMI-002
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
Keywords: Mild Probable Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DBS On (Experimental): DBS system On
  Interventions: Device: DBS-f On
- DBS Off (Sham Comparator): DBS System Off
  Interventions: Device: DBS Off

INTERVENTIONS:
Device: DBS-f On — Deep Brain Stimulation of the fornix
  Arms: DBS On
Device: DBS Off — Deep Brain Stimulation of the fornix turned off
  Arms: DBS Off

SUMMARY:
The primary efficacy objective of this study is to test the hypothesis that DBS-f stimulation (ON) will slow cognitive and functional progression of AD, as compared to no stimulation (OFF), by measuring baseline (pre-implantation) to 12-month change in the integrated Alzheimer's disease rating scale (iADRS).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the subject and caregiver.
2. At least 65 years old
3. Probable Alzheimer's disease according to the National Institute of Aging Alzheimer's disease Association criteria.
4. Mild dementia according to the Clinical Dementia Rating (CDR) global rating of 0.5 or 1 at screening.
5. ADAS-cog-11 score of 10-24 inclusive at screening AND baseline (with a score ≥ 4 on ADAS-cog item 1).
6. Confirmation of Alzheimer's disease based on CSF biomarkers.
7. The patient has an available caregiver or other appropriate knowledgeable informant who can reliably report on daily activities and function and signs the informed consent for participation as such.
8. Patient must be a good surgical candidate for placement of a deep brain stimulator as judged by the DBS surgical team.
9. Fluency (oral and written) in the language in which standardized tests will be administered.
10. The patient is either

    1. taking a stable dose of cholinesterase inhibitor (AChEI) medication (donepezil, galantamine, or rivastigmine) for at least 60 days prior to signing the informed consent form OR
    2. the patient has previously had an intolerance/failure to cholinesterase inhibitor medications that can be documented AND there is no intention to modify the dose over the course of the study (NOTE: These medications may NOT be initiated, discontinued or modified during the 12-month control period).

       OR
    3. c) a physician has fully discussed the possibility of prescribing cholinesterase inhibitors and the physician in collaboration with the patient/caregiver have declined trying cholinesterase inhibitors and this discussion and decision are fully documented in the patient's medical records. This discussion occurred during the course of the patient's care, and not as a component of enrollment or discussion of participation in this clinical trial.

AND there is no intention to modify the dose over the course of the study (NOTE: These medications may NOT be initiated, discontinued or modified after study initiation for the 12-months control period).

Exclusion Criteria:

1. NPI total score ≥ 10 or score ≥ 4 in any NPI domain (clinically significant neuropsychiatric symptoms). Apathy score ≥ 4 acceptable.
2. Modified Hachinski ischemia scale score > 4 at screening.
3. At risk for suicide in the opinion of the investigator or the subject answers "yes" to "Suicidal Ideation" Item 4 or 5 on the C-SSRS (at the time of evaluation) at the screening visit or attempted suicide within the last 2 years.
4. Suffers from a major psychiatric disorder such as schizophrenia, bipolar disorder or major depressive disorder, or has current alcohol or substance abuse based on psychiatric consultation at screening visit.
5. History of moderate or more severe traumatic brain injury in the 2 years prior to signing the consent to participate in the study.
6. History of brain tumor, subdural hematoma, or other clinically significant (in the judgment of the investigator) space-occupying lesion on CT or MRI.
7. History of seizure disorder.
8. Contraindications for MRI scanning, including implanted metallic devices (e.g. non-MRI-safe cardiac pacemaker or neurostimulator; some artificial joints metal pins; surgical clips; or other implanted metal parts), or claustrophobia or discomfort in confined spaces.
9. Radiation exposure in the 1 year prior to signing the informed consent form that, in combination with the radiation exposure from this study, would exceed 5 rem.
10. Abnormal cardiovascular or neurovascular disorder that, in the opinion of the investigator would preclude participation in the study.
11. Currently prescribed or planning to start any amyloid-beta directed antibody drug (e.g. aducanumab or similar) within the first year following implantation in this study. Prior use of amyloid-beta directed antibody drugs must be stopped at least 6 months prior to signing consent.
12. Currently prescribed any non-AD medications that, in the opinion of the investigator would preclude participation in the study.
13. Is unable or unwilling to comply with protocol follow-up requirements.
14. Has a life expectancy of < 1 year.
15. Is actively enrolled in another concurrent clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Over Time at 12 months on the Ingegrated Alzheimer's Disease Rating Scale (iADRS) [ Time Frame: From Baseline to month 12 ] | 12 months
  The iADRS is a composite tool that combines scores from the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) and the Alzheimer's Disease Cooperative Study - instrumental Activities of Daily Living (ADCS-iADL). It measures both cognition and function and demonstrates acceptable psychometric properties, and is effective in capturing both disease progression and separation of placebo and active treatment effect. The iADRS score ranges from 0 to 146 with lower scores indicating worse performance.

SECONDARY OUTCOMES:
Change From Baseline Over Time at 12 months on the Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) [ Time Frame: From Baseline to month 12 ] | 12 months
  The CDR-SB is a validated clinical assessment of global function in patients with AD. Impairment is scored in each of 6 cognitive categories on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2, and severe = 3. The 6 individual category ratings, or "box scores", can be added together to give the CDR-SB which ranges from 0 to 18 (severe impairment).

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas, Austin, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
- Toronto Western Hospital, Toronto, Ontario, Canada
- Germany (7):
  - Universitätmedizin Charité Berlin, Berlin
  - Universitätklinikum Köln, Cologne
  - Universitätsklinikum Schleswig Holstein Campus, Kiel
  - Universität Magdeburg, Magdeburg
  - Technische Universität München, Munich
  - Universitätsklinikum München: Klinik und Poliklinik für Psychiatrie und Psychotherapie Alzheimer Therapie- und Forschungszentrum, München
  - Universitätklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No